CLINICAL TRIAL: NCT00438230
Title: Residual Vein Thrombosis (RVT) Establishes the Optimal Duration of Oral Anticoagulants After a First Episode of Deep Vein Thrombosis of the Lower Limbs
Brief Title: Residual Vein Thrombosis Establishes the Optimal Duration of Oral Anticoagulants
Acronym: DACUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000743
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2007-02-22 (Estimated); Status verified 2007-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Residual vein thrombosis; Optimal duration; Oral anticoagulants
MeSH Terms: conditions — Venous Thrombosis | interventions — Warfarin

INTERVENTIONS:
Drug: Warfarin

SUMMARY:
ABSTRACT Background The optimal duration of oral anticoagulant treatment in patients with idiopathic venous thromboembolism is still uncertain . The present study addressed the possible role of the Residual Vein Thrombosis in assessing the need for a prolonged anticoagulation.

Methods Patients with a first episode of symptomatic unprovoked or provoked proximal Vein Thrombosis (VT) were given Oral Anticoagulant Treatment (OAT) for 3 months. Residual Vein Thrombosis (RVT), ultrasonographically-detected, will be then assessed. Patients without RVT did not continue OAT, whereas those with RVT will be randomized to either stop or continue OAT for 9 more months. Patients were followed-up prospectively focusing on the study outcomes: occurrence of recurrent venous thromboembolism and major bleeding over a period of at least 12 months after OAT discontinuation.

DETAILED DESCRIPTION:
INTRODUCTION Long-term anticoagulant treatment with adjusted doses of vitamin K antagonists is highly effective in preventing recurrent events after a first episode of unprovoked Venous ThromboEmbolism (VTE), even if the optimal duration of this therapy is still uncertain. Since the risk of recurrency is greatest in the first year after the initial thrombotic episode and gradually diminishes thereafter, the benefit of an extended course of anticoagulant treatment may be offset over time by the persisting risk of clinically important bleeding.

A potential clinically relevant approach for establishing the optimal duration of Oral AntCoagulant Therapy (OAT) is that of predicting the individual risk for thrombotic recurrency after the index Deep Vein Thrombosis (DVT). Although the current scheme for establishing the duration of OAT is based on the nature of index DVT (idiopathic or provoked), some new data starting to select other parameters to optimize this decision. Recently, the use of D-dimer has been proven to be effective for selecting OAC duration; however, this investigation evaluated only patients with idiopathic DVT and, moreover, the use of D-dimer can not be easily handle by most of Institutions.

In earlier prospective studies conducted in patients with symptomatic DVT, the presence of a residual thrombus was associated with an increased risk of thrombotic recurrencies either in idiopathic or provoked venous thrombosis. Interestingly, recurrent events occurred not only in the previously affected veins but also in other sites, thus suggesting that Residual Vein Thrombosis (RVT) may express a pro-thrombotic status. Based on these findings, the detection of RVT may be, therefore, of help in establishing the duration of anticoagulation.

To test this hypothesis, we planned a randomized, prospective, follow-up study in patients with a first episode of symptomatic DVT treated with OAT for 3 months. Patients without RVT will not continue anticoagulation, whereas those with RVT will be randomized to either stop or resume anticoagulation.

METHODS Study patients. Patients with a first episode of documented unprovoked and provoked proximal DVT will be eligible for the study if they had completed at least three months of OAT (target INR 2.5, range 2.0-3.0). Provoked DVTs are defined as thrombotic episodes associated with pregnancy or puerperium, recent (i.e. within three months) fracture or plaster casting of a leg, immobilization with confinement to bed for three consecutive days and surgery with general anesthesia lasting longer than 30 minutes. Unprovoked DVTs are defined as thrombotic episodes occurred in apparently healthy individuals. Patients with active cancer, limited life expectancy, antiphospholipid antibody syndrome, or an other known thrombophilic status (such as antithrombin deficiency), serious liver disease, renal insufficiency (serum creatinine > 2 mg/dL), those who lived too far from the center will be excluded from the study. The study has been approved by the institutional review boards of all participating centers. All enrolled patients will provide written informed consent.

Study Design. This is a multicenter prospective study in patients with a first episode of symptomatic (either provoked or idiopathic) proximal DVT detected by Compression UltraSonography (C-US) and receiving OAT [warfarin (Coumadin, Bristol Myers Squibb) for 3 months. At this time, subjects who agreed to participate in the study have a physical examination to assess baseline clinical conditions and to exclude contraindications. C-US of the proximal deep vein system in both legs will be performed, measuring the diameters of any detectable thrombus in the Common Femoral Vein (CFV) and Popliteal Veins (PV). Images will be obtained in transverse section only. Lumen compressibility will be then evaluated on CFV and PV by gentle pressure of the probe, as previously described. Briefly, the major and the minor diameters of the vein segment are measured and recorded before and after compression. C-US findings are scored as "absence of RVT" when residual thrombus occupied, at maximum compressibility, less than 40% of the vein area. Patients without RVT will not continue anticoagulation, whereas those with RVT will be randomized to either stop or continue OAT (INR 2.0-3.0) for additional 9 months. A different randomization sequence for each different study site is computer generated and encapsulated in a randomization computer program. The sequences are balanced by blocks of ten.

Study outcomes and Follow-up. From the assignment visit, patients will be followed up for at least one year after OAT discontinuation; during the follow-up period, patients will be contacted by the clinical centers every 3 months. C-US will be performed only when recurrent symptomatic DVT is suspected. The study outcome is the composite of confirmed recurrent venous thromboembolism (including DVT and/or fatal or non-fatal pulmonary embolism) and major bleeding events from the index DVT to the last day of follow-up. In cases of suspected DVT recurrence the results of ultrasonography will be compared with the previous examination. A diagnosis of recurrent venous thrombosis is made if a previously fully compressible segment (contralateral or ipsilateral) became incompressible. In absence of a previous normal C-US, DVT recurrence is diagnosed if a previously non-occlusive thrombus shifted to occlusive thrombus, provided the vein area before compression had increased by more than 50%); in undetermined cases, contrast venography was performed. In patients with suspected pulmonary embolism, diagnosis of recurrence is based on objective algorithms using clinical probability, ventilation-perfusion lung scanning/helical computed tomography, compression ultrasonography and/or D-dimer if indicated. The diagnosis of clinically relevant haemorrhage will be made in case of decrease of haemoglobin levels > 2.0 gr/dl, retroperitoneal, intracranial or life-threatening. Patients has been instructed to contact the clinical center immediately if symptoms developed suggestive of venous thromboembolism or bleeding. All suspected outcome events and all deaths will be evaluated by a central adjudication committee whose members were unaware of the name of the subject, the enrolling center, the C-US findings and the assigned group.

Statistical analysis. Baseline differences between groups will be assessed by the chi-square test (Yates' correction) for categorical variables and t-test or Mann-Withney U test for continuous variables, as appropriate. Data will be analyzed on intention-to-treat basis. Kaplan-Meier survival curves are plotted to estimate the cumulative incidence of symptomatic recurrent venous thromboembolism and major bleeding. Patients who during the study will develop clinical conditions interfering with the study outcomes (such as ischemic heart disease, cancer, stroke, superficial vein thrombosis, etc) and left the assigned group will be regularly followed-up and included in analysis. Hazard ratios and their 95 percent confidence intervals will be calculated using the Cox's proportional hazards model. The data will be analyzed using the Prism statistical software package (Version 3.0, GraphPad Software Incorporated, San Diego, CA) and the SPSS statistical package (Version 14.0, SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* First episode of unprovoked and provoked proximal DVT of the lower limbs and treated for 3 month with oral anticoagulants

Exclusion Criteria:

* Active cancer,
* Limited life expectancy,
* Antiphospholipid antibody syndrome, or an other known thrombophilic status (such as antithrombin deficiency),
* Serious liver disease,
* Renal insufficiency (serum creatinine > 2 mg/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2003-11; Study Completion 2006-09

PRIMARY OUTCOMES:
Recurrent Venous Thromboembolism
major and minor haemorrhage
death

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Siragusa, MD, Study Chair — University Hospital of Palermo

REFERENCES:
- [Derived] Siragusa S, Malato A, Anastasio R, Cigna V, Milio G, Amato C, Bellisi M, Attanzio MT, Cormaci O, Pellegrino M, Dolce A, Casuccio A, Bajardi G, Mariani G. Residual vein thrombosis to establish duration of anticoagulation after a first episode of deep vein thrombosis: the Duration of Anticoagulation based on Compression UltraSonography (DACUS) study. Blood. 2008 Aug 1;112(3):511-5. doi: 10.1182/blood-2008-01-131656. Epub 2008 May 22. PMID 18497320